CLINICAL TRIAL: NCT03026335
Title: Childhood Resiliency Effects for School-wide Treatment in Belize City
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11403
Record Dates: First submitted 2017-01-06; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Child Behavior
Keywords: Positive Youth Development
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Action Curriculum (Experimental): A school-wide program was implemented in the experimental schools referred to as "Positive Action" and was integrated with the existing Health and Family Life Education curriculum.
  Interventions: Behavioral: Positive Action
- Control/Comparison Group (Active Comparator): Business as usual with students in non-intervened schools
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Positive Action — Based upon a Cognitive Behavioral Therapy model, intervened schools were engaged in providing curriculum, school infrastructure elements, and parent/community involvement activities around a single model aimed to provide positive support for behaviors. Six areas were identified: self-concept, body/mind, responsible self-management, treating others they way you want to be treated, telling yourself the truth, and continual improvement of self.
  Arms: Positive Action Curriculum
Behavioral: Control — Business as usual with students in non-itervened schools
  Arms: Control/Comparison Group

SUMMARY:
The purpose of the study is to use existing school resources and improve identification, referral and local support for children that exhibit exposure to childhood trauma resulting from environmental violence in Belize City. The Ministry of Education has identified the goals of the project to reduce violent behaviors in primary school children and supporting those children that have been exposed to violence or other malicious behavior that would inhibit normal school functioning. In addition, the MOE is supporting additional resources and data collection for a comprehensive evaluation of student behavior and academic performance.

DETAILED DESCRIPTION:
Belize is a country with a developing economy based primarily on agriculture and tourism. Crime and violence are emerging as a threat to the country's governance and business climate. The number of homicides in Belize have increased by more than 30% from 2003-2006. This notion of violence, in particular gang violence, is extremely concerning because the population of Belize is very young. Almost half of the population of Belize is under the age of 18. The youth of Belize are becoming engaged in criminal and delinquent behaviors at an early age that have both individual and societal consequences.

In addition to the violence rates among youth in Belize there is also an educational crisis that must be addressed. Education in Belize is compulsory between the ages of 5-14 and in 2001 93% of 5-14 year old children attended school. Although primary school is mandatory (up to age 14), only about 75% of youth complete primary school and only 25% graduate from secondary school. With few students completing high school it is likely that many may turn to gang related and other illegal activities if they are not prepared to undertake better job opportunities, have not been provided with environmental assets that protect from involvement in risky behavior, and if they are exposed to community/family values that condone gang activity. A number of studies have demonstrated that school-based interventions have moderate effects in reducing violence (average of d = .20 across studies). Combining a sound school-based intervention in Belize that is primarily targeted toward students and teachers, but combined with school-based community/family components designed to heighten awareness of the necessity of protective assets, implemented with local and international support teams, and that fosters positive norms may enhance the effects.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in primary schools under the authority of the Belize Ministry of Education in the Belize District
* Enrolled in eight grades referred to as Infant 1 and 2 (generally aged 5 and 6 years), and 1st through 6th Standard (comprising ages 7 - 12 years)

Exclusion Criteria:

* None

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6296 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Social-Emotional and Character Development Scale | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  28 item self-report scale. A sum of item responses yields an overall score and sub scale scores for self-control, pro-social behavior, respect for teachers, respect for parents, honesty, and self-development. Higher scores represent improved functioning. Scores may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Peer Affiliation Scale | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  7 item self-report scale. A sum of item responses yields a score ranging from 5 to 35 with higher scores representing greater affiliation with peers. Scores may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Behavior Assessment for Children (BASC) | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  6 item sub scale from the BASC comprising a self-report for Anxiety, with higher scores indicting behaviors representative of anxious thought. Scores may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Substance Use and Violent Tendencies Scale | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  Adapted from a CDC measure, this self-report scale contains 11 items that when summed, higher scores represent greater substance use and participation in violence. Scores may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Belief in Moral Center Scale | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  An 11 item self-report measure where higher scores represent belief or adherence to social morality. Item responses are summed, and scores may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Self-Report Scale of Rewards for Pro-Social Behavior | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  A 6 item self-report measure recording how much of the time Parents and Teachers notice when the respondent is nice to others. Item responses are recorded on a 4-point scale. A sum of item responses yield summary scores and may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
School Self-Esteem Scale | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  A 4 item self-report measure asking students how they feel about themselves with respect to school and schoolwork. Item responses are recorded on a 4-point scale. A sum of item responses yield summary scores and may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.
Neighborhood Youth Inventory | Nine (9) months from the beginning of the school year until the end of the school year to coincide with treatment
  A 9 item self-report measure about experiences of the respondent in their neighborhood. Item responses are recorded on a 4-point scale. A sum of item responses yield summary scores and may be reported as raw, percentiles, t-scores, or normal curve equivalent scores.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell M Hull, Ph.D., Principal Investigator — University of North Texas Health Science Center

IPD SHARING:
Plan to Share IPD: No